CLINICAL TRIAL: NCT05676801
Title: Effects of Photodynamic Therapy on the Human Inguinal Skin Microbiome to Improve Antiseptic Effect - Pilot 3
Brief Title: Effect of Photodynamic Therapy on Skin Microbiome. Single Center Study (PHOMIC-III)
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2022_PHOMIC-III
Record Dates: First submitted 2022-12-22; First posted 2023-01-09 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Prosthesis and Implants; Surgical Site Infection; Prosthetic Joint Infection; Postoperative Wound Infection Deep Incisional Surgical Site
MeSH Terms: conditions — Surgical Wound Infection | interventions — Photochemotherapy

STUDY DESIGN:
Intervention Model Description: All patients get Photodynamic treatment in addition to skin antisepsis. (The contrallateral side of the leg is our control side, therefore only one arm)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PDT group (Experimental): PDT with 5% topical methyl aminolevulinate (MAL) before skin antisepsis
  Interventions: Drug: Photodynamic Therapy

INTERVENTIONS:
Drug: Photodynamic Therapy — PDT with methyl aminolevulinate (MAL) as the prodrug for the photosensitizer Pp IX

SUMMARY:
The overarching aim of this research project is to prevent orthopedic implant-associated infections. This study aims to investigate if PDT has an effect on bacterial skin colonization in order to improve skin antisepsis strategies for the prevention of surgical site infections.

DETAILED DESCRIPTION:
Periprosthetic joint infections are a feared complication after orthopedic surgery in particular in our increasing elderly population. These infections are usually difficult to treat, because microorganisms persist in biofilms on the orthopedic implant surface. Therefore, it would be desirable to prevent these infections. It is hypothesized that bacteria from the skin surface or dermis - such as Staphylococcus aureus, coagulase-negative staphylococci, or Cutibacterium sp. - are transmitted into the periimplant tissue during surgery. In an interdisciplinary study with the Orthopedic University Hospital Balgrist, the investigators see that common skin antisepsis preparation is not effective to eliminate skin bacteria before surgery because they might persist in sebaceous or sweat glands. Photodynamic therapy (PDT) has the potential to improve skin antisepsis as we recently showed. The PDT works here on the one hand through a long-lasting destruction of the sebaceous glands, and on the other hand due to anti-inflammatory and bactericidal effects.

In a previous pilot study, the investigators tested if skin antisepsis can be improved with previous PDT using the photosensitizer-inducing prodrug 5% topical methyl aminolevulinate (MAL) on inguinal skin in 10 healthy participants. The induced photosensitizer was protoporphyrin IX (Pp IX) activated by red light (633 nm). The investigators showed 100% killing of colonizing skin bacteria at the same day after this treatment. However, orthopedic surgeons are hesitant to perform an arthroplasty surgery after such a treatment due to the side effects of skin erythema for a few days.

In a follow up study, the investigators tested the PDT effect using 5-aminolevulinic acid (5-ALA) induced Pp IX with a daylight lamp (400-750nm) and achieved 70% skin sterility with skin redness only in a minority of participants. The sterilizing effect lasted up to 3 days.

The investigators are entirely convinced about this novel prevention concept using daylight but need to identify the photosensitizer with the ideal balance of bactericidal effect versus skin irritation. Building upon the gathered data, the investigators will explore PDT with longer incubation time of the photosensitizer MAL and the less toxic and pain free illumination with daylight.

Primary outcome:

Effect of photodynamic therapy with the photosensitizer Pp IX (MAL) and daylight in combination with surgical skin antisepsis on bacterial skin colonization on the day of application and on day 3 after PDT.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female participants ≥ 18 years who volunteer for the pilot study, in which a routine photodynamic treatment at the Department of Dermatology will be performed and effect of skin colonization will be analyzed, and who signed an informed consent (after information about the project)

Exclusion Criteria:

* Pregnant and breastfeeding women
* Participants with inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc.,
* Participants taking antibiotics in the 14 days prior to PDT or until follow-up at 21 days
* Participants who received oral retinoid therapy within the last 6 months
* Participants who received anti-inflammatory agents as Non-Steroidal Anti-Inflammatory Drugs (NSAIDs) within the 14 days prior and after the PDT
* Participants taking any photosensitizing drugs within 4 weeks prior to PDT
* Participants who had a history of photosensitivity disorder
* Fitzpatrick's skin phototype V-VI

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-02-04 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Culture results of skin swabs | within 10 days after PDT
  Quantitative evaluation of bacterial density and species from skin swabs taken before PDT, immediately after PDT, and after after skin antisepsis using culture technique

CONTACTS AND LOCATIONS:
Overall Officials: Yvonne Achermann, PD Dr. med., Principal Investigator — Dermatology
Locations (1):
- University Hospital of Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided